CLINICAL TRIAL: NCT06463379
Title: The Efficacy of Intravenous Pulse in Attaining Remission in Refractory Juvenile Idiopathic Arthritis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mahrous, Professor, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00000049
Record Dates: First submitted 2024-06-01; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Refractory Juvenile Idiopathic Arthritis (Despite 2 DMARDs Still Active)
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pulse steroid (Experimental): 108 patients will receive 125 mg solumedrol intravenous pulse for 2 consecutive days plus their concomitant medication.
  Interventions: Drug: Solumedrol
- without pulse (Placebo Comparator): 107 patients will not receive any additional medications.
  Interventions: Drug: Solumedrol

INTERVENTIONS:
Drug: Solumedrol — 2 days pulse steroid injection 125 mg methylrednisolone

SUMMARY:
Interventional phase 3 study aiming to unravel the value of pulse steroids in achieving remission or low disease activity in refractory active JIA

DETAILED DESCRIPTION:
First group will receive 2 consecutive days intravenous pulse of 125 mg methylprednisolone.

Second group will not receive additional drugs. Assessment was done at baseline and every month for 3 months for both groups using Juvenile Arthritis Disease Activity Score (JADAS) and the American College of Rheumatology Pediatric 30, 50, and 70 response criteria (ACR Pedi. 30, 50, 70).

ELIGIBILITY:
Inclusion Criteria:

* Patients still active despite administration o 2 DMARDs

Exclusion Criteria:

* Other connective tissue diseases
* Endocrine disorders such as Thyroid disorders.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 215 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
remission or low disease activity | 3 months
  patients will be assessed at baseline and every month for 3 months using Juvenile Arthritis Disease Activity Score (JADAS) for disease activity American College of Rheumatology Pediatric 30, 50, and 70 (ACR Pedi. 30, 50, 70) for disease activity

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No